CLINICAL TRIAL: NCT02778880
Title: A Randomized Controlled Trial of Intranasal Sub-dissociative Dosing of Ketamine Compared to Intranasal Fentanyl for Treatment of Pain Associated With Acute Extremity Injuries in Children
Brief Title: Pain Reduction With Intranasal Medications for Extremity Injuries
Acronym: PRIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN_PRIME_001
Record Dates: First submitted 2016-04-19; First posted 2016-05-20 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2018-10

CONDITIONS: Pain; Traumatic Limb Injury
MeSH Terms: conditions — Pain | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Ketamine 1.5 mg/kg intranasally for one dose
  Interventions: Drug: Ketamine
- Fentanyl (Active Comparator): Fentanyl 2 mcg/kg intranasally for one dose
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine
  Other Names: Ketalar
  Arms: Ketamine
Drug: Fentanyl
  Arms: Fentanyl

SUMMARY:
This study compares the analgesic effect of intranasal sub-dissociative dosing of ketamine and intranasal fentanyl in children presenting to the Emergency Department with acute extremity injuries.

DETAILED DESCRIPTION:
Inadequate pain control, especially in the emergency department (ED), is a major public health concern. Despite increased awareness, pain continues to be underdiagnosed and undertreated, particularly in the pediatric population. Children often encounter long delays in medication administration, possibly due to the time required to obtain intravenous access. The intranasal administration route offers a more efficient alternative for faster and noninvasive delivery of pain medication. This route is gaining popularity secondary to its rapid onset of active, minimal discomfort and relative simplicity.

Opioids are the most commonly used class of analgesic pain medication for children presenting in severe pain due to traumatic injuries. Despite their potential effectiveness, opioids have several concerning adverse effects, particularly when administered prior to procedural sedation in children. Administration of pre-procedural sedation opioids is associated with an increased risk of serious adverse events (oxygen desaturation, apnea, and hypotension) as well as the need for significant interventions, such as bag-mask ventilation, intubation, and pharmacologic blood pressure support. In addition, due to genetic variations that may lead to increased or diminished opioid sensitivity, ideal dosing to adequately control severe pain yet avoid adverse medication-related side effects is difficult to ascertain. Many children in severe pain do not receive opioids, receive doses that are below those recommended or experience long delays in receiving opioids. The reasons for this are unclear, but the investigators speculate that this may be due in part to fear of adverse effects of opioids, provider inexperience with opioid use in children or fear of contributing to opioid tolerance or abuse. For all of these reasons, providers often seek non-opioid alternatives for pediatric patients with acute, severe pain.

Ketamine, in sub-dissociative doses administered by the intravenous or intranasal route, is emerging as an alternative medication for the treatment of moderate to severe pain in multiple settings. In adults, low dose ketamine is well tolerated and has been used successfully as an adjuvant and an alternative to opioids to provide rapid pain relief in the ED. As a dissociative anesthetic, ketamine is the most commonly used agent to facilitate painful procedures in the pediatric emergency department. At lower doses, it has been used in children to provide analgesia in a variety of acute and chronic pain settings, including terminal diagnoses, sickle cell disease, perioperative pain, traumatic injuries, extensive burns and conditions where opioids are contraindicated. Similar to adults, ketamine has been used via the intranasal route to provide adequate analgesia and sedation in children in the pre-hospital setting and in those undergoing procedures.

The objective of this study is to compare intranasal sub-dissociative ketamine with intranasal fentanyl for treatment of acute pain associated with traumatic limb injuries in children presenting to the ED and to document an objective respiratory side effect profile utilizing noninvasive capnometry. If found to be an effective analgesic, intranasal ketamine would be particularly useful in children who experience adverse effects with opioids, have developed opioid tolerance as a result of chronic painful conditions, have poor opioid sensitivity due to their genetic predisposition or in pediatric trauma patients with the potential for hypotension. Additionally, for patients that require procedural sedation for fracture reduction, avoiding opioids early in the emergency department visit may decrease sedation recovery time and the risk of serious adverse events during sedation.

ELIGIBILITY:
Inclusion Criteria:

* 8 years to 17 years (up to the 18th birthday)
* Presenting to emergency department with one or more extremity injuries
* Visual analog scale score 35 mm or greater
* Parent or legal guardian present and willing to provide written consent

Exclusion Criteria:

* Received narcotic pain medication prior to arrival
* Evidence of significant head, chest, abdomen, or spine injury
* Glasgow coma score less than 15 or unable to self report pain score
* Nasal trauma or aberrant nasal/airway anatomy
* Active epistaxis
* Allergy to ketamine, fentanyl or meperidine
* Non-English speaking parent and/or child
* History of psychosis
* Postmenarchal female without a urine or serum assay documenting the absence of pregnancy
* Brought in my juvenile detention center or in police custody
* Pregnancy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa M Frey, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Matthew R Mittiga, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frey TM, Florin TA, Caruso M, Zhang N, Zhang Y, Mittiga MR. Effect of Intranasal Ketamine vs Fentanyl on Pain Reduction for Extremity Injuries in Children: The PRIME Randomized Clinical Trial. JAMA Pediatr. 2019 Feb 1;173(2):140-146. doi: 10.1001/jamapediatrics.2018.4582. PMID 30592476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This clinical trial took place at a tertiary care children's hospital emergency department from March 2016 to February 2017. The study sample was identified through an established triage process identifying children with an acute painful extremity injury. These patients were ages 8-17 years with a visual analog scale (VAS) score greater than 35 mm.
Period: Overall Study
Arm/Group | Ketamine | Fentanyl
Started | 45 | 45
Completed | 44 | 42
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Fentanyl | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (2.6) | 12.2 (2.3) | 12.0 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 26 | 31 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 30 | 29 | 59
  Race/Ethnicity: Black | 11 | 10 | 21
  Race/Ethnicity: Hispanic | 0 | 2 | 2
  Race/Ethnicity: Other | 3 | 1 | 4
Weight [Mean (Standard Deviation); unit: kilograms] | 45.8 (14.4) | 50.8 (22.8) | 48.3 (18.6)
Mechanism of Injury [Count of Participants; unit: Participants]
  Sports Related/Recreational | 30 | 26 | 56
  Motor Vehicle Accident | 1 | 2 | 3
  Fall | 10 | 13 | 23
  Other | 3 | 1 | 4
Time of injury prior to arrival [Median (Inter-Quartile Range); unit: minutes] | 43.0 [27.0 to 63.0] | 51.5 [30.0 to 85.0] | 47.3 [28.5 to 74.0]
Extremity [Number; unit: participants] — Three participants had more than one extremity involved. Therefore, percentages do not add up to 100.
  participants
    Upper Extremity | 33 | 28 | 61
    Lower Extremity | 13 | 15 | 28
Diagnosis [Number; unit: participants] — Two participants had both a fracture and a dislocation.
  participants
    Fracture | 39 | 34 | 73
    Dislocation | 4 | 2 | 6
    Sprain/Strain | 1 | 5 | 6
    Other | 2 | 1 | 3
Reduction Required [Count of Participants; unit: Participants] | 19 | 23 | 42
Sedation Required [Count of Participants; unit: Participants] | 19 | 20 | 39
Analgesic Prior to Arrival [Count of Participants; unit: Participants]
  Ibuprofen | 4 | 4 | 8
  Acetaminophen | 1 | 2 | 3
  Naproxen | 0 | 1 | 1
  No Analgesic | 39 | 35 | 74
Initial VAS score [Mean (Standard Deviation); unit: score on a scale] — The Visual Analog Scale is a pain scale ranging from 0 mm (no pain) to 100 mm (worst possible pain) that has been shown to be valid and reliable in children 8 to 17 years of age suffering from acute pain. A minimum clinically significant difference in VAS score ranges from 10 to 12 mm. in children and adolescents. The optimal cut off points between mild, moderate, and severe pain are 35 mm and 60 mm. Population: One patient in the Ketamine group did not have a baseline pain score documented.
  score on a scale
    number analyzed (Participants) | 43 | 42 | 85
    (all) | 74.7 (15.3) | 72.0 (18.6) | 73.4 (17.0)
Baseline Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 90.8 (15.2) | 88.6 (14.8) | 89.7 (15.0)
Baseline Respiratory Rate [Mean (Standard Deviation); unit: breaths per minute] | 22.1 (6.6) | 23.0 (7.4) | 22.5 (7.0)
Baseline Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 126.5 (19.1) | 128.9 (19.6) | 127.7 (19.4)
Baseline Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.9 (13.6) | 73.5 (12.9) | 76.3 (13.5)
Baseline Oxygen Saturation [Mean (Standard Deviation); unit: percent] | 99.8 (0.6) | 99.6 (0.6) | 99.7 (0.6)
Baseline End Tidal Captometry [Mean (Standard Deviation); unit: mmHg] | 36.6 (6.4) | 38.0 (4.4) | 37.3 (5.5)
Time to Study Medication from Arrival [Mean (Standard Deviation); unit: minutes] | 26.6 (9.9) | 26.1 (10.3) | 26.4 (10.1)
Volume of Study Medication Administered [Median (Inter-Quartile Range); unit: milliliters] | 1.3 [1.1 to 1.6] | 1.8 [1.3 to 2.0] | 1.6 [1.2 to 1.8]
Dose of Study Medication Administered (Ketamine) [Median (Inter-Quartile Range); unit: milligrams per kilogram (mg/kg)] — Population: Participants receiving Fentanyl did not receive Ketamine
  milligrams per kilogram (mg/kg)
    number analyzed (Participants) | 44 | 0 | 44
    (all) | 1.5 [1.5 to 1.5] |  | 1.5 [1.5 to 1.5]
Dose of Study Medication Administered (Fentanyl) [Median (Inter-Quartile Range); unit: micrograms per kilogram (mcg/kg)] — Population: Participants receiving Ketamine did not receive Fentanyl
  micrograms per kilogram (mcg/kg)
    number analyzed (Participants) | 0 | 42 | 42
    (all) |  | 1.9 [1.7 to 1.9] | 1.9 [1.7 to 1.9]

OUTCOME MEASURES:

1. Primary Outcome: Difference From Baseline in Visual Analog Scale Pain Score
Description: A VAS score is a self reported pain score of 0-100 millimeters (0 = no pain; 100 = worst possible pain). A decrease in a VAS score indicates a decrease in pain severity.
Time Frame: 30 minutes after study medication
Population: One patient in the ketamine group did not have a baseline pain score documented and four patients withdrew from the study (1 in the ketamine group, 3 in the fentanyl group), resulting in 43 patients randomized to the ketamine group and 42 patients randomized to the fentanyl group included in the primary outcome analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 43 | 42
score on a scale | -30.6 [-35.8 to -25.4] | -31.9 [-37.2 to -26.6]

2. Secondary Outcome: Difference From Baseline in Visual Analog Scale Pain Score
Description: as for outcome 1
Time Frame: 15 minutes after study medication
Population: One patient in the ketamine group did not have a baseline pain score documented and four patients withdrew from the study (1 in the ketamine group, 3 in the fentanyl group), resulting in 43 patients randomized to the ketamine group and 42 patients randomized to the fentanyl group included in this secondary outcome analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 43 | 42
score on a scale | -24.4 [-29.3 to -19.4] | -25.3 [-30.3 to -20.3]

3. Secondary Outcome: Difference From Baseline in Visual Analog Scale Pain Score
Description: as for outcome 1
Time Frame: 60 minutes after study medication
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
score on a scale | -27.7 [-33.8 to -21.6] | -29.0 [-35.1 to -22.8]

4. Secondary Outcome: Highest Achieved University of Michigan Sedation Scale (UMSS) Score
Description: The University of Michigan Sedation Scale is a valid and reliable tool that allows for rapid assessment of the depth of sedation in children. It is a simple observational tool that assesses the level of alertness on a five-point scale. It has been validated in children and has shown to have significant inter-rater reliability. Score is 0-4 (0 = awake and alert; 1= minimally sedated; 2 = moderately sedated; 3 = deeply sedated; 4 = unarousable)
Time Frame: 15, 30, and 60 minutes after study medication administration
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
Participants
  UMSS 0 | 23 | 32
  UMSS 1 | 17 | 9
  UMSS 2 | 4 | 1

5. Secondary Outcome: Rescue Analgesia
Description: Documentation of additional pain medication after study medication administration
Time Frame: Within the first 60 minutes after study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
Participants
  Ibuprofen | 1 | 3
  Fentanyl | 1 | 3
  Morphine | 7 | 3
  Ketamine | 1 | 0
  Toradol | 1 | 0
  No rescue analgesia | 33 | 33

6. Secondary Outcome: Heart Rate
Time Frame: 15 minutes after study medication
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
beats per minute | 90.1 (12.8) | 84.4 (14.1)

7. Secondary Outcome: Heart Rate
Time Frame: 30 minutes after study medication
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
beats per minute | 90.5 (12.8) | 85.6 (13.5)

8. Secondary Outcome: Heart Rate
Time Frame: 60 minutes after study medication
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
beats per minute | 85.1 (12.4) | 82.9 (12.9)

9. Secondary Outcome: Respiratory Rate
Time Frame: 15 minutes after study medication
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
breaths per minute | 23.1 (11.9) | 22.3 (5.8)

10. Secondary Outcome: Respiratory Rate
Time Frame: 30 minutes after study medication
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
breaths per minute | 23.3 (8.7) | 19.9 (5.7)

11. Secondary Outcome: Respiratory Rate
Time Frame: 60 minutes after study medication
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
breaths per minute | 21.8 (8.1) | 19.7 (5.7)

12. Secondary Outcome: Systolic Blood Pressure
Time Frame: 15 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 127.3 (18.0) | 127.9 (19.3)

13. Secondary Outcome: Systolic Blood Pressure
Time Frame: 30 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 126.3 (15.0) | 123.4 (15.6)

14. Secondary Outcome: Systolic Blood Pressure
Time Frame: 60 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 122.3 (14.9) | 122.0 (15.1)

15. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 15 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 76.1 (10.7) | 73.4 (12.7)

16. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 30 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 76.3 (10.3) | 73.6 (11.2)

17. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 60 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 70.8 (9.2) | 70.6 (10.4)

18. Secondary Outcome: Oxygen Saturation
Time Frame: 15 minutes after study medication
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
percent | 99.6 (0.7) | 99.2 (0.9)

19. Secondary Outcome: Oxygen Saturation
Time Frame: 30 minutes after study medication
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
percent | 99.5 (0.7) | 99.4 (0.9)

20. Secondary Outcome: Oxygen Saturation
Time Frame: 60 minutes after study medication
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
percent | 99.3 (0.9) | 99.3 (0.9)

21. Secondary Outcome: Capnometry Value
Time Frame: 15 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 36.6 (5.2) | 38.3 (4.2)

22. Secondary Outcome: Capnometry Value
Time Frame: 30 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 38.6 (5.6) | 40.4 (6.8)

23. Secondary Outcome: Capnometry Value
Time Frame: 60 minutes after study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 44 | 42
mmHg | 38.7 (4.2) | 38.9 (5.4)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ketamine | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42
Other Adverse Events (participants affected / at risk) | 34/44 | 13/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=44) | Fentanyl (N=42)
Dizziness (Nervous system disorders) | 9 | 7
Dysphoria/Dissociation (Nervous system disorders) | 1 | 0
Unpleasant Taste (Gastrointestinal disorders) | 9 | 2
Drowsiness (Nervous system disorders) | 21 | 10
Nausea/Vomiting (Gastrointestinal disorders) | 3 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Vision Changes (Eye disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Lightheadedness (Nervous system disorders) | 2 | 0
Nystagmus (Eye disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Convenience sample; 4 patients withdrew before medication given; Conservative choice of non-inferiority margin; Interventions like splinting or child life presence were not assessed; Rescue analgesia was at the discretion of the primary provider

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT02778880/Prot_SAP_000.pdf